CLINICAL TRIAL: NCT01978925
Title: Effectiveness Pharmaceutical Care at Discharge in the Emergency Department: a Randomized Controlled Trial
Brief Title: Pharmaceutical Care in Emergency Department
Acronym: AMPaRAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Moinhos de Vento (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMPaRAR 01
Record Dates: First submitted 2013-11-01; First posted 2013-11-08 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Medication Adherence; Hypertension; Diabetes Mellitus
Keywords: Pharmaceutical care; Medication Adherence; Blood Pressure; Diabetes; Emergency
MeSH Terms: conditions — Medication Adherence; Hypertension; Diabetes Mellitus; Emergencies | interventions — Pharmaceutical Services

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pharmaceutical care (Experimental): In the ED, immediately after discharge, participants randomized to the pharmaceutical care group will receive intervention coordinated by the study pharmacist.
  Interventions: Other: Pharmaceutical care
- Usual care (No Intervention): In addition to counseling provided by a physician and by the nursing staff during their stay in the ED (usual care), patients randomized to the control group will receive the same printed material information on hypertension and/or diabetes medications and lifestyle interventions in order to keep patients masked.

INTERVENTIONS:
Other: Pharmaceutical care — The clinical pharmacist will provide a structured 30-minute intervention for enhancing their medication adherence.
  The recommendations include: discussion on hypertension and/or diabetes, risk of complications, prescribed drug therapy, correct use of medications and proper dosage, possible adverse effects, route of administration, schedule of administration and correct storage. The pharmacist will also emphasize the importance of lifestyle modifications. Printed educational material, with information on hypertension and/ or diabetes medications, including suggested lifestyle interventions was prepared to assist in the intervention and will be handed to patients in the end of the session.
  Arms: Pharmaceutical care

SUMMARY:
The purpose of this study is to evaluate the effectiveness of pharmaceutical care, compared to usual care, in patient discharge in an emergency department in patients with hypertension and/or diabetes mellitus type 2.

DETAILED DESCRIPTION:
This is a randomized controlled, single-center study, with blinding of outcome assessors. A pilot study with ten patients was previously conducted in order to test study logistics and data collection instruments. Participants will be recruited from a public ED at Restinga district in Porto Alegre, southern Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Blood pressure inadequate control (systolic blood pressure ≥ 160 or diastolic blood pressure ≥ 100 mmHg) or
* Diabetes mellitus inadequate Control( ≥ 200 mg/dL) or hypoglycemia moderate or severe
* Be referred to clinical care.

Exclusion Criteria:

* < 18 years
* Not resident of Porto Alegre
* Diabetes mellitus type I
* Unable to answer the questionnaire or to sign the informed consent form
* Hospital admission
* Death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Medication Adherence | Two months
  Outcome of interest: High Adherence According to the Brief Medication Questionnaire and Morisky-Green Test

SECONDARY OUTCOMES:
Blood Pressure Control | Two months
Glycated hemoglobin (HbA1C) for diabetic patients | two months
Quality of Life | Two months

OTHER OUTCOMES:
Fasting plasma glucose for diabetic patients | Two months

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo A Ribeiro, PhD, Principal Investigator — Hospital Moinhos de Vento
Locations (1):
- Emergency Department - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Kuhmmer R, Lima KM, Ribeiro RA, Hammes LS, Bastos GA, Cotta de Souza MC, Polanczyk CA, Soares Rollin GA, Caon S, Guterres CM, Araujo Leite LE, Delabary TS, Falavigna M. Effectiveness of pharmaceutical care at discharge in the emergency department: study protocol of a randomized controlled trial. Trials. 2015 Feb 25;16:60. doi: 10.1186/s13063-015-0579-3. PMID 25888343